CLINICAL TRIAL: NCT06574802
Title: Combined Application of Er:YAG Laser and Sub-gingival Air Polishing Powder in Treatment of Periodontitis: A Split-mouth, Randomized Controlled Trial
Brief Title: Er:YAG Laser and Air Polishing Application in Periodontal Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CYFH202207
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-08

CONDITIONS: Periodontitis
Keywords: generalized, stage Ⅱ or stage Ⅲ
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Active Comparator): Er:YAG laser (ERL) plus sub-gingival air polishing treatment
  Interventions: Procedure: ERL + air polishing
- control group (Placebo Comparator): ERL treatment only
  Interventions: Procedure: ERL

INTERVENTIONS:
Procedure: ERL + air polishing — Er:YAG laser (ERL) plus sub-gingival air polishing treatment
  Arms: test group
Procedure: ERL — ERL treatment
  Arms: control group

SUMMARY:
Periodontitis (gum disease) is an infection of the gums that can lead to tooth loss. In recent years, many types of dental lasers or other devices have been used for the non-surgical treatment of periodontal diseases. However, it remains unclear whether the combined application of laser and air polishing is effective as an adjuvant treatment for periodontitis. The purpose of this study is to compare the use of combined application of Er:YAG laser and sub-gingival air polishing powder, with the treatment of Er:YAG laser only, in periodontal diseases treatment in a Chinese population.

DETAILED DESCRIPTION:
The study will use a split-mouth design, two quadrants (one quadrant from each jaw) were randomly allocated to either the test or control group. The quadrants in the test group received Er:YAG laser (ERL) plus sub-gingival air polishing treatment, while the quadrants in the control group received ERL only. Clinical periodontal examinations were evaluated at baseline, 3 months, 6 months, 1 year, and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* 1) aged 35-65 years old, in good systemic healthy;
* 2) clinically diagnosed with generalized stage Ⅱ or stage Ⅲ periodontitis;
* 3) a minimum of 20 teeth

Exclusion Criteria:

* 1) pregnancy or recent pregnancy plans;
* 2) had received periodontal treatment within the previous 6 months;
* 3) taken antibiotics within the previous 3 months;
* 4) had diabetes;
* 5) obvious malocclusion, history of orthodontic treatment, or a habit of mouth breathing.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Changes in PD | at 3 months, 6 months, 1 year, and 2 years
  Changes in probing depth (PD) measured using periodontal probing
Changes in CAL | at 3 months, 6 months, 1 year, and 2 years
  Changes in clinical attachment level (CAL) measured using periodontal probing

SECONDARY OUTCOMES:
changes in BI | at 3 months, 6 months, 1 year, and 2 years
  Changes in bleeding index (BI) measured using periodontal probing
PLI | at 3 months, 6 months, 1 year, and 2 years
  Plaque index (PLI) assessed by an examiner using a scale of 0 to 3

CONTACTS AND LOCATIONS:
Overall Officials: GuangXu Liu, Doctor, Principal Investigator — Research Department
Locations (1):
- Beijing Chao Yang Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No